CLINICAL TRIAL: NCT02687529
Title: Evaluation of the 4th Generation QuantiFERON-TB Test (QFT-Plus) for the Detection of Tuberculosis Infection
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CST001_USA7
Record Dates: First submitted 2016-02-16; First posted 2016-02-22 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low Risk: Tested with CST001
  Interventions: Device: CST001
- Known Risk: Tested with CST001
  Interventions: Device: CST001

INTERVENTIONS:
Device: CST001

SUMMARY:
To compare the positivity rate of the investigational assay to the currently approved QuantiFERON-TB Gold In-Tube assay.

ELIGIBILITY:
Low Risk and Known Risk Cohorts

Inclusion Criteria:

* Compensated and uncompensated members (current or future) of the Department of Veterans Affairs with no identified symptoms of active TB disease
* Age greater than 18 years or less than 80 years.

Exclusion Criteria:

* Currently taking therapy for active tuberculosis or latent TB infection for more than 14 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have either a low risk or known risk for TB exposure.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2015-11-07 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System (VAPAHCS), Palo Alto, California, United States

REFERENCES:
- [Background] QuantiFERON-TB Gold Package Insert (DOC. No. US05990301L). March 2013. QIAGEN Inc.
- [Background] Shams H, Klucar P, Weis SE, Lalvani A, Moonan PK, Safi H, Wizel B, Ewer K, Nepom GT, Lewinsohn DM, Andersen P, Barnes PF. Characterization of a Mycobacterium tuberculosis peptide that is recognized by human CD4+ and CD8+ T cells in the context of multiple HLA alleles. J Immunol. 2004 Aug 1;173(3):1966-77. doi: 10.4049/jimmunol.173.3.1966. PMID 15265931
- [Background] Lewinsohn DA, Winata E, Swarbrick GM, Tanner KE, Cook MS, Null MD, Cansler ME, Sette A, Sidney J, Lewinsohn DM. Immunodominant tuberculosis CD8 antigens preferentially restricted by HLA-B. PLoS Pathog. 2007 Sep 21;3(9):1240-9. doi: 10.1371/journal.ppat.0030127. PMID 17892322

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Risk; Known Risk: Tested with CST001
  CST001
Period: Overall Study
Arm/Group | Low Risk | Known Risk
Started | 34 | 32
Completed | 34 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk | Known Risk | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 29 | 60
  >=65 years | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 52.5 [24 to 68] | 58.5 [26 to 67] | 55.5 [24 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 23 | 16 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 32 | 29 | 61
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 22 | 29
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 6 | 4 | 10
  White | 18 | 5 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Concordant CST001 Assay Results for All Replicates Across Three Testing Sites
Description: To demonstrate the reproducibility of the CST001 assay between 3 external laboratories with 2 operators per site.
Time Frame: 1 day (At time of enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk | Known Risk
Number analyzed (Participants) | 34 | 32
Participants | 32 | 23
Statistical Analysis 1: Comparison: Low Risk vs Known Risk; Test type: Equivalence — The number of positive and negative CST001 assay results for each subject, across all sites and operators were compared. In order for a subject to have a concordant result, the same assay call must be observed for all replicates across all sites (6/6); proportion of concordant calls = 83.33, 95% CI 2-sided [72.13 to 91.38]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Low Risk | Known Risk
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 0/34 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No